CLINICAL TRIAL: NCT03961334
Title: MidregiOnal Proatrial Natriuretic Peptide to Guide SEcondary Stroke Prevention: The MOSES-study. An International, Multicentre, Randomised-controlled, Two-arm, Assessor-blinded Trial
Brief Title: MidregiOnal Proatrial Natriuretic Peptide to Guide SEcondary Stroke Prevention
Acronym: MOSES
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Mira Katan, Prof. Dr. med., University of Zurich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MOSES
Record Dates: First submitted 2019-05-16; First posted 2019-05-23 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke | interventions — Dabigatran; apixaban; edoxaban; Aspirin; Clopidogrel

STUDY DESIGN:
Masking Description: Blinded endpoint assessment by independent CEC
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DOACs (Experimental): Direct oral anticoagulants
  Interventions: Drug: Dabigatran; Drug: Apixaban; Drug: Edoxaban
- Antiplatelets (Active Comparator): SOC therapy with antiplatelets until study completion or until detection of AF. After detection of AF treatment with DOAC becomes SOC.
  Interventions: Drug: Aspirin; Drug: Clopidogrel

INTERVENTIONS:
Drug: Dabigatran — 150mg 2x/d
  Other Names: Pradaxa
  Arms: DOACs
Drug: Apixaban — 5mg 2x/d
  Other Names: Eliquis
  Arms: DOACs
Drug: Edoxaban — 60mg 1x/d
  Other Names: Lixiana
  Arms: DOACs
Drug: Aspirin — 100mg 1x/d
  Other Names: Aspirin cardio
  Arms: Antiplatelets
Drug: Clopidogrel — 75mg 1x/d
  Arms: Antiplatelets

SUMMARY:
The present trial is addressing the question if a biologically distinct subgroup of ischemic stroke patients without known atrial fibrillation at admission, selected by a cut-off level of MRproANP concentration, which represents a underlying increased risk of cardiac thrombogenicity, benefits from direct oral anticoagulation (DOAC) within 7 days of symptom onset versus standard of care (antiplatelet) as preventive treatment.

DETAILED DESCRIPTION:
Three DOACs with marketing authorisation in Switzerland and the EU for the prevention of stroke and systemic embolism in patients with atrial fibrillation can be used. Eligible patients will be randomly assigned to either the standard of care (control) or the experimental (direct start with DOAC) arm with a ratio of 1:1. Each study participant will be observed during a follow up period within one year after index stroke.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ischemic stroke
* level ≥200pmol/L within 72 hours from symptom onset
* Age ≥ 18 years
* Signed informed consent

Exclusion Criteria:

* History of AF, AF on 12-lead ECG on admission or any AF ≥30 seconds during heart-rhythm monitoring prior to randomization
* Other condition that require anticoagulant therapy (e.g., venous thromboembolism) as per Investigator's judgment including therapeutical dose of low-molecular-weight heparin or heparin
* Strong likelihood to be treated with prolonged (i.e. more than 30 days) dual antiplatelet therapy during the course of the trial (such as coronary stenting, etc.)
* Patients undergoing planned procedures where therapy with a DOAC is a contraindication (e.g. surgery)
* Previous intracranial hemorrhage in the last year
* Evidence of severe cerebral amyloid angiopathy if MRI scan performed
* Chronic kidney disease with creatinin clearance <30ml/min and or subject who requires haemodialysis or peritoneal dialysis
* Known bleeding diathesis (e.g. active peptic ulcer disease , platelet count < 100'000/mm3 or haemoglobin < 9 g/dl or INR ≥ 1.7, documented haemorrhagic tendencies or blood dyscrasias)
* Active infective endocarditis
* CT or MRI evidence of cerebral vasculitis
* Known allergy or intolerance to antiplatelets or DOACs
* Female who is pregnant or lactating or has a positive pregnancy test at time of admission
* Current participation in another drug trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2019-12-05 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Recurrent stroke of any type | within one year after index stroke
  The primary outcome measure is the time to any recurrent stroke (ischemic, hemorrhagic, unspecified, or fatal stroke)

SECONDARY OUTCOMES:
Composite of major bleeding, recurrent stroke and/or vascular death | within one year after index stroke
  Composite of major bleeding, recurrent stroke and/or vascular death (whichever occurs first)
Major bleeding, recurrent stroke and/or vascular death as single components | within one year after index stroke
  Each single component of the composite in outcome 2 (major bleeding, recurrent stroke and/or vascular death)

CONTACTS AND LOCATIONS:
Overall Officials: Mira Katan, Prof.Dr.med., Principal Investigator — University Hospital, Basel, Switzerland
Locations (14):
- Attikon University Hospital, Athens, Greece
- Oslo University Hospital - Ullevål, Oslo, Norway
- Spain (3):
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario Virgen Macarena, Seville
  - Campus Hospital Universitario Virgen del Rocío, Seville
- Switzerland (8):
  - Kantonsspital Aarau, Department of Neurology, Aarau, Canton of Aargau
  - University Hospital of Basel, Basel
  - University Hospital of Bern/Inselspital, Bern
  - Ospedale Regionale di Lugano, Ente Ospedaliero Cantonale, Lugano
  - Kantonsspital St.Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - Klinik Hirslanden, Zurich
  - University Hospital of Zurich, Department of Neurology, Zurich
- Queen Elizabeth University Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No